CLINICAL TRIAL: NCT01502072
Title: An Open Label Randomized Controlled Trial To Prevent the Progression of Respiratory Syncytial Virus Upper Respiratory Tract Infection to Lower Respiratory Tract Infection in Patients After Hematopoietic Stem Cell Transplant
Brief Title: Respiratory Syncytial Virus - RSV Protocol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0813; NCI-2012-00021 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-12-22; First posted 2011-12-30 (Estimated); Results first posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-01

CONDITIONS: Bone Marrow Transplant Infection; Infection in Marrow Transplant Recipients; Respiratory Syncytial Virus Infections; Respiratory Syncytial Virus Pneumonia; Cancer; Acute Leukemia
Keywords: Ribavirin; Ribavirin Aerosol; Respiratory Syncytial Virus; RSV; upper respiratory tract infection; URI; Lower respiratory tract Infection; LRI; pneumonia; aerosolized ribavirin; HSCT; Hematopoietic stem cell transplantation; oral ribavirin therapy
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Neoplasms; Respiratory Tract Infections; Pneumonia | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Inhaled Ribavirin (Experimental): Group 1: Inhaled form of Ribavirin 60 milligrams/milliliter 3 times/day for 3 hours for up to 10 days.
  Interventions: Drug: Ribavirin
- Oral Ribavirin (Experimental): Group 2: Ribavirin Capsules 20 mg/kg orally 3 times/day for up to 10 days.
  Interventions: Drug: Ribavirin
- No Ribavirin (No Intervention): Group 3: No Ribavirin treatment.

INTERVENTIONS:
Drug: Ribavirin — Modified schedule of 60 milligrams/milliliter for 3-hour period 3 times/day for at least 5 days by aerosolization via a SPAG-2 generator via a face mask.
  Arms: Inhaled Ribavirin
Drug: Ribavirin — One time loading dose of 10 mg/kg oral dose then 20 mg/kg orally (rounded to the nearest 200 mg dose) divided into three doses per day (max 1800 mg/day).
  Arms: Oral Ribavirin

SUMMARY:
The goal of this clinical research study is to learn if ribavirin can help to control RSV in patients with immune systems that have been weakened by a stem cell transplant. Researchers also want to compare the effectiveness of the drug when it is given by mouth to when it is inhaled. The safety of the drug in both methods of delivery will be studied.

Ribavirin is designed to prevent the RSV virus from making more copies of itself in the body.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study and the study doctor thinks that the disease requires treatment at this time, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups. You will have an equal chance of being assigned to either group:

* If you are in Group 1, you will receive the inhaled form of ribavirin. You will inhale ribavirin 3 times a day for 3 hours each time in a tent in a hospital room. You will receive the drug for up to 10 days.
* If you are in Group 2, you will take capsules of ribavirin 3 times a day for up to 10 days.

If the study doctor does not think that the disease requires treatment at this time, you will be assigned to Group 3. If you are in Group 3, you will not receive treatment with ribavirin, but you will have the same tests and procedures at the study visits described below.

Study Visits:

At all study visits, you will be asked about how you are feeling, about any side effects or symptoms you may be having, and about any other drugs you may be taking.

On Day 3 (+/- 1 day):

* You will have a physical exam, including measurement of your vital signs
* Your nasal passages will be checked for RSV.

On Days 7 and 14 (+/- 1 day):

* Blood (about 2 teaspoons) will be drawn for routine tests.
* You will have a physical exam, including measurement of your vital signs
* Your nasal passages will be checked for RSV.

Length of Study:

If you are in Groups 1 or 2, you will receive the study drug for up to 10 days. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions. If your doctor thinks you need treatment longer than 10 days, you will receive that as part of your routine care. This may mean changing to receiving the drug in inhaled form if you began the study receiving it by mouth.

All participants will have end-of-study and follow-up visits, as described below.

End-of-Study Visit:

If you are in Groups 1 or 2, the end-of-study visit will be about 14 days after your last dose of the study drug. If you are in Group 3, the end-of-study visit will take place at about Day 21. The following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs.
* Blood (about 4 teaspoons) will be drawn for routine tests and to check for RSV antibodies.
* Your nasal passages will be checked for RSV.
* You will be asked about how you are feeling, about any side effects or symptoms you may be having, and about any drugs you may be taking.

Follow-Up Visit:

About 6 to 10 weeks after your last dose of study drug, you will have a pulmonary function test to check your lung function.

This is an investigational study. Ribavirin is FDA approved and commercially available for the treatment of hepatitis C when given by mouth, and for severe RSV in children when inhaled. Giving the drug to adults with weak immune systems after a stem cell transplant is investigational.

Up to 96 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. HSCT patients with either moderate or severe immunodeficiency based on immunodeficiency scoring system would be eligible for entry on study if a nasopharyngeal wash or throat swab specimen is positive by rapid RSV antigen testing and/or on culture within 72 hours (therapeutic arms). (Please see Appendix E for definitions and Immunodeficiency Scoring).
2. HSCT patients with mild immunodeficiency based on immunodeficiency scoring system would be eligible for entry on study if a nasopharyngeal wash or throat swab specimen is positive by rapid RSV antigen testing and/or on culture within 72 hours but will not be randomized to therapeutic arms and will be followed as per standard of care (control arm).
3. Patients must be at least 18 years of age and able to swallow pills.
4. Patients with RSV infection limited to the URT as documented by negative Chest radiographic findings within the last 48 hours of enrollment and pulse oxygenation of more than 90 mm of Hg on room air.
5. Women of child bearing potential with a negative urine or blood pregnancy test within a month of enrollment (only for patients who are going to be randomised to either therapeutic arms).
6. Patients with Hemoglobin levels more than or equal to 8 g/dl would be eligible for the study even if they are currently receiving blood products.
7. Patients may receive up to 2 doses of aerosolized ribavirin (modified regimen) before enrollment into the study.
8. Patients who will be enrolled on the observational arm should meet inclusion criteria # 2, 3, and 4 only.

Exclusion Criteria:

1. Patients with previous history of hypersensitivity to ribavirin or its components
2. Women who are pregnant or plan a pregnancy within 8 weeks after completion of treatment (only for patients who are going to be randomised to either therapeutic arms).
3. Patients with evidence of RSV LRI as documented by a positive rapid RSV antigen testing and/or culture on nasal washes AND new or progressive infiltrates on chest radiographic studies suggestive of viral etiology and/or pulse oxygen less than 90 mm of Hg on room air.
4. Patients with positive RSV by rapid antigen testing and/or culture in bronchoalveolar lavage regardless of the chest radiographic findings.
5. Patients who are considered to be moderately or severely anemic as per the NCI classification will not be included in the study, i.e patients with hemoglobin level less than 8 g/dl
6. Patient with Total Bilirubin and Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) three times the upper limit of normal.
7. Male partners of women who are pregnant (only for patients who are going to be randomised to either therapeutic arms).
8. Patients with known history of autoimmune hepatitis, Hepatitic C or those with hemoglobinopathies (eg, thalassemia major, sickle cell anemia).
9. Patients with creatinine clearance of less than or equal to 50 ml/Min
10. Patients taking didanosine, azathioprine, or nucleoside reverse transcriptase inhibitors
11. Patients who will be enrolled on the observational arm should not meet exclusion criteria #3 and 4 only.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-12-28 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy F. Chemaly, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: December 2011 - March 2016. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: 48 participants enrolled, 4 participants did not meet enrollment criteria after screening labs were performed.
Groups:
- Oral Ribavirin: Ribavirin Capsules 20 mg/kg orally 3 times/day for up to 10 days.
  Ribavirin: One time loading dose of 10 mg/kg oral dose then 20 mg/kg orally (rounded to the nearest 200 mg dose) divided into three doses per day (max 1800 mg/day).
- Inhaled Ribavirin: Inhaled form of Ribavirin 60 milligrams/milliliter 3 times/day for 3 hours for up to 10 days.
- No Ribavirin: No Ribavirin treatment.
Period: Overall Study
Arm/Group | Oral Ribavirin | Inhaled Ribavirin | No Ribavirin
Started | 14 | 10 | 20
Completed | 13 | 9 | 20
Not Completed | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Death | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: One patient from the Oral ribavarin group withdrew consent.
Groups:
- Oral Ribavirin: Ribavirin Capsules 20 mg/kg orally 3 times/day for up to 10 days.
- Total: Total of all reporting groups
Arm/Group | Oral Ribavirin | Inhaled Ribavirin | No Ribavirin | Total
Number analyzed (Participants) | 13 | 10 | 20 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (9.9) | 58.2 (12.6) | 41.5 (17.1) | 50.8 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 12 | 22
  Male | 7 | 6 | 8 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 7 | 11
  Not Hispanic or Latino | 12 | 7 | 13 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 3 | 4
  White | 11 | 7 | 8 | 26
  More than one race | 1 | 3 | 7 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 10 | 20 | 43

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression to Lower Respiratory Tract Infection (LRI)
Description: Patient who developed signs of lower respiratory tract infection
Time Frame: 14 days
Measure: Number; unit: percentage of participants
Arm/Group | Oral Ribavirin | Inhaled Ribavirin | No Ribavirin
Number analyzed (Participants) | 13 | 10 | 20
percentage of participants | 8 | 30 | 10

ADVERSE EVENTS:
Time Frame: At baseline, up to 2 weeks
Arm/Group | Oral Ribavirin | Inhaled Ribavirin | No Ribavirin
All-Cause Mortality (participants affected / at risk) | 0/13 | 1/10 | 0/20
Serious Adverse Events (participants affected / at risk) | 3/13 | 5/10 | 5/20
Other Adverse Events (participants affected / at risk) | 4/13 | 4/10 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Ribavirin (N=13) | Inhaled Ribavirin (N=10) | No Ribavirin (N=20)
Altered mental status (Psychiatric disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 3
Graft versus host disease (General disorders) | 0 | 0 | 1
Acute renal failure (Renal and urinary disorders) | 0 | 1 | 0
Alveolar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
GI bleed (Gastrointestinal disorders) | 1 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Ribavirin (N=13) | Inhaled Ribavirin (N=10) | No Ribavirin (N=20)
Worsening oral ulcer (Ear and labyrinth disorders) | 1 | 0 | 0
Shortness of breath/hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Clausterphobia (Psychiatric disorders) | 0 | 1 | 0
Seizure (Psychiatric disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Jitteriness (Psychiatric disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT01502072/Prot_SAP_000.pdf